CLINICAL TRIAL: NCT06232109
Title: Phase 1, Open-Label, Parallel Group Drug-Drug Interaction Study to Assess the Effect of Fluvoxamine (CYP2C19 Inhibitor), Itraconazole (CYP3A4 Inhibitor) and Paroxetine (CYP2D6 Inhibitor) on the Pharmacokinetics of ASN51 in Healthy Subjects
Brief Title: Drug-Drug Interaction of ASN51 With Fluvoxamine, Itraconazole and Paroxetine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asceneuron S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASN51-104
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — Fluvoxamine; Itraconazole; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASN51 (No Intervention)
- ASN51 + Fluvoxamine (Experimental)
  Interventions: Drug: Fluvoxamine; Drug: ASN51
- ASN51 + Itraconazole (Experimental)
  Interventions: Drug: Itraconazole; Drug: ASN51
- ASN51 + Paroxetine (Experimental)
  Interventions: Drug: Paroxetine; Drug: ASN51

INTERVENTIONS:
Drug: Fluvoxamine — Oral
  Arms: ASN51 + Fluvoxamine
Drug: Itraconazole — Oral
  Arms: ASN51 + Itraconazole
Drug: Paroxetine — Oral
  Arms: ASN51 + Paroxetine
Drug: ASN51 — Oral
  Arms: ASN51 + Fluvoxamine; ASN51 + Itraconazole; ASN51 + Paroxetine

SUMMARY:
The drug-drug interaction study has been designed to investigate the effect of Fluvoxamine, Itraconazole and Paroxetine on the pharmacokinetics of ASN51

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males or females of nonchildbearing potential
* Aged 18-55 years (inclusive) at time of Screening
* Deemed healthy based on medical history, physical and neurological examination, electrocardiogram (ECG), vital signs, and laboratory tests of blood and urine
* Body weight ≥ 50.0 kg (men) or ≥ 45.0 kg (women) at Screening
* Body mass index (BMI); Quetelet index in the range 18.0-30.9 kg/m2 (inclusive) at Screening

Key Exclusion Criteria:

* Clinically relevant abnormal medical history, physical or neurological findings, ECG, or laboratory values at Screening, or before the first dose of any study medication, that could interfere with the objectives of the study or the safety of the subject
* History or presence of acute or chronic illness, or clinically-significant medical abnormality, sufficient to invalidate the subject's participation in the study or make it unnecessarily hazardous
* History or presence of any disease, medical condition, or surgery (e.g., stomach bypass), likely to affect the absorption, distribution, metabolism, or excretion of medicines. Subjects with a history of cholecystectomy
* Presence or history of severe or clinically significant adverse reaction to any drug; or a history of sensitivity to ASN51 (all subjects), or any components of the medications
* Receipt of an investigational product or device within 6 weeks (or 5 half-lives, or twice the duration of the biological effect, of the investigational product, if known - whichever is longer) before the first dose of study medication; in the follow-up period of another clinical study at the time of Screening for this study
* Use of a prescription medicine during the 14 days (or 5 half-lives of the medicine, if known - whichever is longer) before the first dose of study medication
* Use of an over-the-counter medicine, including vitamins, herbal, or dietary supplements (including St John's Wort), with the exception of acetaminophen (paracetamol), during the 7 days (or 5 half-lives of the medicine, if known - whichever is longer, or 28 days if the medicine is a potential hepatic enzyme inducer) before the first dose of study medication
* Positive test for hepatitis B, hepatitis C or human immunodeficiency virus (HIV)

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Cmax of ASN51 | Up to Day 15
Tmax of ASN51 | Up to Day 15
AUC0-tau of ASN51 | Up to Day 15
AUC0-inf of ASN51 | Up to Day 15
t1/2 of ASN51 | Up to Day 15
λz of ASN51 | Up to Day 15

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Pokorny, MD, Study Chair — Asceneuron, SA; Jeroen v Wetering, MD, Principal Investigator — QPS Holdings LLC
Locations (1):
- ICON Groningen Van Swietenlaan 6, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No